CLINICAL TRIAL: NCT00634309
Title: Candesartan Cilexetil in Heart Failure Assessment of Reduction in Mortality and Morbidity. Clinical Study of Candesartan in Patients With Heart Failure and Depressed Left Ventricular Systolic Function
Brief Title: Candesartan Cilexetil in Heart Failure Assessment of Reduction in Mortality and Morbidity (CHARM Added)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH-AHS-0006; D2454C00006
Record Dates: First submitted 2008-03-07; First posted 2008-03-13 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Atacand; Candesartan
MeSH Terms: conditions — Heart Failure | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Candesartan
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Candesartan
  Other Names: Atacand
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
A study to evaluate the effect of Atacand on patients with heart failure with depressed left ventricular function

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or above
* Congestive Heart Failure with symptoms for more than 4 weeks before starting study
* Provision of informed consent

Exclusion Criteria:

* Current low blood pressure with symptoms
* Liver disease considered significant by the study doctor
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Estimated)
Dates: Start 1999-06; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality or hospitalisation due to congestive heart failure | 2, 4, 6 weeks, 6 months, every 4 months thereafter until 24 months

SECONDARY OUTCOMES:
Cardiovascular mortality or hospitalisation for management of congestive heart failure, or non fatal MI | 2, 4, 6 weeks, 6 months, every 4 months thereafter until 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. JJV McMurray, Principal Investigator

REFERENCES:
- [Derived] Kondo T, Dewan P, Anand IS, Desai AS, Packer M, Zile MR, Pfeffer MA, Solomon SD, Abraham WT, Shah SJ, Lam CSP, Jhund PS, McMurray JJV. Clinical Characteristics and Outcomes in Patients With Heart Failure: Are There Thresholds and Inflection Points in Left Ventricular Ejection Fraction and Thresholds Justifying a Clinical Classification? Circulation. 2023 Aug 29;148(9):732-749. doi: 10.1161/CIRCULATIONAHA.122.063642. Epub 2023 Jun 27. PMID 37366061
- [Derived] Lund LH, Claggett B, Liu J, Lam CS, Jhund PS, Rosano GM, Swedberg K, Yusuf S, Granger CB, Pfeffer MA, McMurray JJV, Solomon SD. Heart failure with mid-range ejection fraction in CHARM: characteristics, outcomes and effect of candesartan across the entire ejection fraction spectrum. Eur J Heart Fail. 2018 Aug;20(8):1230-1239. doi: 10.1002/ejhf.1149. Epub 2018 Feb 12. PMID 29431256
- [Derived] Desai AS, Claggett B, Pfeffer MA, Bello N, Finn PV, Granger CB, McMurray JJ, Pocock S, Swedberg K, Yusuf S, Solomon SD. Influence of hospitalization for cardiovascular versus noncardiovascular reasons on subsequent mortality in patients with chronic heart failure across the spectrum of ejection fraction. Circ Heart Fail. 2014 Nov;7(6):895-902. doi: 10.1161/CIRCHEARTFAILURE.114.001567. Epub 2014 Oct 17. PMID 25326006
- [Derived] Preiss D, Zetterstrand S, McMurray JJ, Ostergren J, Michelson EL, Granger CB, Yusuf S, Swedberg K, Pfeffer MA, Gerstein HC, Sattar N; Candesartan in Heart Failure Assessment of Reduction in Mortality and Morbidity Investigators. Predictors of development of diabetes in patients with chronic heart failure in the Candesartan in Heart Failure Assessment of Reduction in Mortality and Morbidity (CHARM) program. Diabetes Care. 2009 May;32(5):915-20. doi: 10.2337/dc08-1709. Epub 2009 Feb 5. PMID 19196892